CLINICAL TRIAL: NCT07001280
Title: Garadacimab Real-world Treatment Outcomes of Effectiveness, Safety, and Quality-of-Life in Patients With HAE (GREAT Study)
Brief Title: A Study Investigating the Effectiveness and Safety of Garadacimab for Treating Patients With Hereditary Angioedema (HAE)
Acronym: GREAT
Status: Recruiting | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CSL312_4001
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedemas
Keywords: Angioedema; Genetic disorder; Long term prophylaxis; Health-related quality of life
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Garadacimab: This cohort will include all participants diagnosed with HAE and who will be prescribed garadacimab treatment as per routine clinical practice.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be administered as part of this study.

SUMMARY:
This is a multinational, multicenter, prospective, observational cohort study of patients with HAE in the real-world setting. The study will include patients newly initiating garadacimab in routine clinical practice. Each participant will be followed for 48 months after index date (date of the first administration of garadacimab).

Patient data will be collected from the HAE eDiary, patient medical records (MRs) and/or during a routine clinical visit and will be entered into the electronic case report form (eCRF) via an electronic data capture (EDC) system. Data pertaining to HAE attacks, prior HAE treatments, retrospective focused safety data collection, and healthcare resource utilization (HCRU) over a look-back period of 12 months prior to the enrollment will be extracted from the MR, and patients will also record retrospective HAE attack related data over a look-back period of 3 months prior to enrollment in the HAE eDiary.

The primary aim of this study is to investigate the real-world effectiveness of garadacimab as measured by HAE attack rate before and after garadacimab initiation in patients with HAE over 24 months of follow-up. The study will aim to complement the data available from the clinical development program on the efficacy, safety, and health-related quality-of-life (HRQoL) in patients with HAE taking garadacimab.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants aged greater than or equal to (>=) 12 years at enrollment.
* 2. Participants with clinical and/or laboratory confirmed diagnosis of HAE.
* 3. Participants newly initiating garadacimab, as prescribed according to the decision of the treating physician per routine clinical practice and in accordance with the indication per the approved local label, independent of and prior to enrollment in the study.
* 4. Willing and able to provide written informed consent and/or assent by parent or legal guardian for children less than (<) 18 years of age (or legal age of consent in the respective countries).
* 5. Ability to use an electronic device such as a smartphone or a computer for data collection in the study.

Exclusion Criteria:

* 1. Participants with a concomitant diagnosis of another form of angioedema such as idiopathic or acquired angioedema, recurrent angioedema associated with urticaria (histaminergic angioedema).
* 2. Participants participating in any ongoing interventional clinical study, including interventional studies with garadacimab. Participants in this study who later chose to enroll in any interventional clinical study (including garadacimab) will be discontinued from this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with the diagnosis of HAE and who will initiate garadacimab treatment per routine clinical practice will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate Ratio (IRR) of HAE Attacks | Up to 24 months
  Monthly HAE attack rate while on treatment with garadacimab, including all HAE attacks, HAE attacks requiring acute treatment (on demand therapy [ODT]), and by severity will be reported. All HAE attacks will be categorized by severity as: Mild (no impact on daily life), Moderate (some impact on daily life), and Severe (severe impact on daily life).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs), Severity of AEs, Serious AEs (SAEs), and Treatment-related AEs | Up to 48 months
Change From Baseline in Angioedema Control Test (AECT) Total Score | Baseline to 48 months
  The AECT includes a set of 4 AECT items attributable to the domains of signs and symptoms, impact and effectiveness of treatment, and the 4th item addresses the important aspect of unpredictability, which correlates strongly with anxiety and fears of recurrent angioedema patients. Score ranges from 0 (minimum) to 16 (maximum). A higher score indicates a higher level of angioedema control.
Change From Baseline in Angioedema Quality of Life Questionnaire (AE-QoL) Total Score | Baseline to 48 months
  The AE-QoL includes 17 items across 4 domains: functioning (4 items), fatigue/mood (5 items), fears/shame (6 items), and food (2 items). Total scores range from 0 to 100, where 100 indicates the worst possible impairment of health related QoL.
Percentage of Participants With Reduction in Monthly HAE Attacks and who Achieved HAE Attack-free Status | Up to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Global Program Director, Study Director — CSL Behring
Locations (9):
- United States (4):
  - Medical Research of Arizona, Phoenix, Arizona
  - John Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Riverside Medical Group, Belleville, Belleville, New Jersey
- Germany (5):
  - HZRM Haemophilie-Zentrum Rhein Main, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Leipzig, Saxony
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Hamburg, Schleswig-Holstein
  - Charité - Campus Charité Mitte, Berlin

IPD SHARING:
Plan to Share IPD: No